CLINICAL TRIAL: NCT01079260
Title: An Investigation of the Efficacy of High Energy, Low Volume Oral Nutritional Supplements in Participants at Risk of Malnutrition
Brief Title: An Investigation of the Efficacy of Oral Nutritional Supplements in Participants at Risk of Malnutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NCC300
Record Dates: First submitted 2010-02-25; First posted 2010-03-03 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Malnutrition
Keywords: Malnourished; Elderly; Nutrition support
MeSH Terms: conditions — Malnutrition | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard ONS (Active Comparator)
  Interventions: Dietary Supplement: Standard ONS
- High Energy, Low volume ONS (Experimental): High energy, low volume ONS
  Interventions: Dietary Supplement: High Energy, low volume ONS

INTERVENTIONS:
Dietary Supplement: Standard ONS — Standard ONS
  Other Names: ONS; sip feeds; Oral nutritional supplements
  Arms: Standard ONS
Dietary Supplement: High Energy, low volume ONS — High energy, low volume ONS
  Other Names: ONS; Sip feeds; Oral nutritional supplements
  Arms: High Energy, Low volume ONS

SUMMARY:
This study aims to investigate the efficacy of high energy, low volume oral nutritional supplements (ONS) compared to equivalent standard ONS (control) to maximize nutrient intake, compliance, gastro intestinal tolerance and function, in participants at risk of malnutrition.

DETAILED DESCRIPTION:
In current clinical practice malnourished (undernourished) patients may receive oral nutritional supplements (ONS) to aid in the management of their malnutrition (undernutrition). Poor compliance to ONS was been reported in the scientific literature, however recent studies of a low volume, high energy ONS have shown high compliance. This study aims to further explore compliance to low volume ONS compared to standard ONS. This study is a 2 week cross over study with a 4 week optional extension. Participants at risk of malnutrition will receive a low volume, high energy ONS for 1 week and a standard ONS for 1 week in a random order to compare nutrient intake and compliance. This short term element of the study was designed based on a similar study by Hubbard et al 2009, where significant differences in compliance and energy intake were observed. Participants may then take part in an optional 4 week extension period where they will receive their preferred ONS for 4 weeks. Longer term outcomes such as change in weight, muscle function and tolerance to the ONS will be measured in this part of the study. Changes in weight and muscle function are typically seen in 4 weeks.

Overview of the study:

1. Participants will be assessed for inclusion and exclusion criteria by the investigating dietitian or research nurse, and then provided with information about the study. Eligible participants will be asked for their written informed consent. Participant characteristics and medical history will be collected.
2. Participants will be randomly allocated to receive either:

A. A standard ONS (1.5kcal/ml) as control, ad libitum in addition to diet for 7 days. Participants will then receive the high energy, low volume equivalent ONS (2.4kcal/ml) ad libitum in addition to diet for 7 days (n=70), or:

B. A high energy, low volume ONS (2.4kcal/ml) ad libitum in addition to diet for 7 days. Participants will then receive the equivalent standard ONS (1.5kcal/ml) as control, ad libitum in addition to diet for 7 days (n=70). Participants will then have an option to continue with their preferred ONS for a further 4 weeks (28 days).

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age > 18 years
* At risk of malnutrition (medium or high risk of malnutrition with 'Malnutrition Universal Screening Tool', 'MUST' score ≥ 1)
* Competent to provide written informed consent and able to answer questions
* No requirement for tube or parenteral feeding
* Willingness to take part in the study and to follow the study protocol

Exclusion Criteria:

* Requirement for tube or parenteral nutrition
* Participants receiving palliative care
* Participants with chronic renal disease requiring dialysis
* Participants with liver failure
* Participants that are pregnant or lactating
* Participation in other studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-02; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Nutrient intake (energy, protein and micronutrients) | 1week
  Dietary intake, including the intake of all foods, drinks and ONS will be recorded at baseline (day 1), at the end of week 1, at the end of week 2 and at the end of the optional extension period (week 6) using 24 hr dietary recall. A dietary analysis program will be used to calculate intake from food and total dietary intake.

SECONDARY OUTCOMES:
Compliance with ONS | 1week
  Participants' compliance with ONS (percentage of bottle consumed), will be recorded on a daily basis by the participant or their carer throughout the study.
ONS Acceptability (taste, aroma) and ONS Preference (which type is preferred) | 1week
  The acceptability (taste, texture, aroma) and preference for the type of ONS will be assessed (using Yes/No questions and visual analogue scales) to gather patients feedback on the acceptability the the supplements
Appetite | 1week
  The effect of the ONS on hunger and fullness will be assessed by questionnaire using visual analogue scales at baseline (day 1), at the end of week 1, at the end of week 2 and at the end of the study (week 6).
Anthropometry | 6weeks
  At baseline as part of screening with MUST, at the end of week 1, at the end of week 2 and at the end of the study (week 6), body weight (kg) will be measured using standard methods and body mass index (kg/m2) calculated. Body weight will be measured to the nearest 0.1kg using a weighing scale or weighing chair without shoes or heavy clothing.
Muscle Strength (Hand Grip Strength) | 6weeks
  Hand grip strength will be measured at baseline (day 1), at the end of week 2 and at the end of the study (week 6) using a handgrip dynamometer.
Gastro-intestinal (GI) tolerance | 6weeks
  Gastro-intestinal tolerance will be assessed at baseline (day 1), at the end of week 1, at the end of week 2 and the end of week 6 for 1 day, using a standardized GI tolerance questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Stratton, Principal Investigator — Nutricia UK Ltd
Locations (1):
- Dietetics Dept, Great Western Hospital, Swindon, Wiltshire, United Kingdom